CLINICAL TRIAL: NCT01063647
Title: Allogeneic Hematopoietic Stem Cell Transplantation in Patients With Advanced Hematological Malignancies After Treosulfan-based Conditioning Therapy - A Clinical Phase II Study
Brief Title: Dose-range Finding Treosulfan-based Conditioning
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: medac GmbH (Industry)
Responsible Party: Joachim Baumgart, PhD, medac GmbH
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MC-FludT.6/L
Record Dates: First submitted 2010-02-03; First posted 2010-02-05 (Estimated); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Hematological Malignancies
Keywords: Treosulfan; Allogeneic stem cell transplantation; Conditioning therapy
MeSH Terms: conditions — Hematologic Neoplasms | interventions — treosulfan

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 1 (Experimental): Treosulfan: 10 g/m² i.v. on 3 consecutive days (day -6 to -4)
  Interventions: Drug: Treosulfan
- 2 (Experimental): Treosulfan:12 g/m² i.v. on 3 consecutive days (day -6 to -4)
  Interventions: Drug: Treosulfan
- 3 (Experimental): Treosulfan: 14 g/m² i.v. on 3 consecutive days (day -6 to -4)
  Interventions: Drug: Treosulfan

INTERVENTIONS:
Drug: Treosulfan — 10 g/m² i.v. infusion, day -6, -5, -4
  Other Names: Ovastat
  Arms: 1
Drug: Treosulfan — 12 g/m² i.v. infusion, day -6, -5, -4
  Other Names: Ovastat
  Arms: 2
Drug: Treosulfan — 14 g/m² i.v. infusion, day -6, -5, -4
  Other Names: Ovastat
  Arms: 3

SUMMARY:
Evaluation of the safety and efficacy of 3 x 10, 3 x 12 or 3 x 14 g/m² Treosulfan resp., combined with 5 x 30 mg/m² fludarabine prior to allogeneic, hematopoietic stem cell transplantation of patients with hematological malignancies, but non-eligible to standard conditioning treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with a haematological chemosensitive malignancy indicated for an allogeneic transplantation, but presenting an increased toxicity risk for classical (high-dose busulfan or standard-dose total body irradiation) conditioning therapies (remission criteria ref. to Appendix L):

   * CML in first or subsequent chronic phase
   * NHL in 2nd CR/PR, chemosensitive PR after autologous transplantation ; CLL in 2nd or subsequent CR/PR
   * Relapsed Morbus Hodgkin (MH) after autologous transplantation
   * Multiple Myeloma (MM) stage II and III according to Durie and Salmon
   * AML in 2nd CR/PR or high-risk AML in 1st CR/PR

   High-risk defined for example by the following:
   * Cytogenetics: -5/5q, -7/7q, del(5q), abnormalities of 3q, complex karyotype (> 3 abnormalities), or
   * PR after 1 cycle of induction therapy
   * ALL in 2nd CR/PR or high-risk ALL in 1st CR/PR

   High-risk defined as follows:
   * Leukocytes > 3000/µl (B-Linage) or > 100000/µl (T-Linage);
   * Pro-B-ALL, pre-T-ALL
   * Cytogenetics: t(9;22)/BCR-ABL; t(4;11)/ALL1-AF
   * MDS (patients without prior chemotherapy may be included)
2. Availability of an HLA-identical sibling donor (MRD) or HLA-identical unrelated donor (MUD) or one mismatch (out of the 6 standard markers) sibling donor (1 misMRD):

   • HLA-identity defined by the following markers: A, B, DRB1. DQB1 must be recorded.
3. Age > 18 years
4. Karnofsky Index > 80 %
5. Adequate contraception in female patients of child-bearing potential
6. Co-operative behavior of individual patients
7. Written informed consent

Exclusion Criteria:

1. Completely chemotherapy-resistant disease
2. Severe cardiac insufficiency, severe cardio-vascular or other severe concomitant diseases
3. Symptomatic malignant involvement of the CNS
4. Active infectious disease
5. HIV-positive or active hepatitis infection
6. Impaired liver function (Bilirubin > 1.5 x upper normal limit; Transaminases > 3.0 x upper normal limit)
7. Impaired renal function (Creatinine-clearance < 60 ml/min; Serum Creatinine > 1.5 x upper normal limit).
8. Pleural effusion or ascites > 1.0 L
9. Pregnancy or lactation
10. Known hypersensitivity to fludarabine and/or treosulfan
11. Parallel participation in another experimental drug trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2001-11; Primary Completion 2005-06 (Actual); Study Completion 2006-06 (Actual)

PRIMARY OUTCOMES:
Safety - Evaluation of feasibility and tolerability of 3 x 10, 12 or 14 g/m² Treosulfan combined with 5 x 30 mg/m² fludarabine prior to allogeneic stem cell transplantation • frequency and severity of TRM until 6 months after transplantation | 6 months

SECONDARY OUTCOMES:
Efficacy - Evaluation of the proportion of relapse- and/or progression free patients six months after transplantation (using standard remission criteria) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Mathias Freund, MD, Principal Investigator — University Hospital Rostock
Locations (7):
- Helsinki University Central Hospital, Helsinki, Finland
- Germany (4):
  - Charité University Hospital Berlin, Berlin
  - University Hospital Hamburg Eppendorf, Hamburg
  - 5th Medical Clinic, Clinic North, Nuremberg
  - University Hospital Rostock, Rostock
- Silesian Medical University, Katowice, Poland
- Karolinska University Hospital & Karolinska Institute, Stockholm, Sweden